CLINICAL TRIAL: NCT00415389
Title: The Stroke Warning Information and Faster Treatment Study (SWIFT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Approval lapse
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AAAA9948; P50NS049060 (NIH)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Stroke
Keywords: Stroke; interactive educational program; acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): interactive educational program
  Interventions: Behavioral: interactive educational program
- 2 (Active Comparator): usual medical care
  Interventions: Behavioral: usual medical care

INTERVENTIONS:
Behavioral: interactive educational program — 2-session interactive stroke educational program
  Arms: 1
Behavioral: usual medical care — standard educational materials and usual care
  Arms: 2

SUMMARY:
The purposes of this study are to determine the effectiveness of an interactive stroke educational program compared to standard educational materials and usual care, to increase stroke knowledge, and to improve emergency room arrival times upon onset of stroke symptoms.

DETAILED DESCRIPTION:
Rapid diagnosis and treatment of acute ischemic stroke is critical to reduce disability and death caused by stroke. While recombinant tissue plasminogen activator, or rt-PA, is the only approved treatment for acute ischemic stroke, less than 2-3 percent of individuals with stroke actually receive treatment. The inability to capture acute ischemic stroke cases within 3 hours of symptom onset is one critical factor. Populations at highest risk for stroke are significantly undereducated about the need for rapid, intervention upon onset of stroke symptoms. This is especially true among vulnerable populations including African Americans, Hispanics, and the poor.

The purpose of this study is to evaluate the effectiveness of a 2-session, culturally-sensitive, interactive stroke educational program compared to standard educational materials and usual care. In this study, the scientists will determine if the interactive program increases knowledge about stroke, and results in earlier arrival to the emergency room in the case of stroke.

The study will enroll 1400 individuals who have had a stroke or transient ischemic attack (TIA). Participants will be randomized to receive usual medical care--which includes standard educational information on stroke, stroke warning signs and risk factors--or usual medical care plus a 2-session interactive stroke educational program. All participants will be administered pre and post (30 days and 1 year) intervention stroke knowledge/behavior surveys. In additional, participants will be contacted every 12 months to check health status and document new stroke events associated with emergency room arrival time.

The SWIFT study is part of the Specialized Program for Translational Research in Acute Stroke (SPOTRIAS), which seeks to understand why certain people may be at increased risk for stroke. The goal of the study is to increase stroke knowledge, change behavior, and improve emergency room arrival times upon onset of stroke symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral infarction/TIA hospitalized at New York Presbyterian Hospital (Milstein Hospital and Allen Pavilion)
* 18 year-old and older at onset of the stroke
* Self-identified as of White, Black or Hispanic race-ethnicity
* Living in a household with a telephone

Exclusion Criteria:

* Patients unable to give informed consent
* Discharged to nursing home or requiring 24 hour care.
* A Modified Rankin score > 4 at baseline
* Severe aphasia or severe cognitive impairment limiting comprehension
* Pre-stroke dementia history
* Patients with end stage cancer, or other medical conditions resulting in mortality </= 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1635 (Actual)
Dates: Start 2005-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Surveillance methodologies will measure arrival times of acute strokes from stroke symptoms onset to ER among participants for the length of the study, as well as increase in stroke knowledge at one month and one year post stroke event. | at one month and one year post stroke event

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Boden-Albala, DrPH, Principal Investigator — Columbia University
Locations (1):
- Neurological Institute, 710 W 168th Street, 6th Floor, Room 640, New York, New York, United States

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Boden-Albala B, Stillman J, Roberts ET, Quarles LW, Glymour MM, Chong J, Moats H, Torrico V, Parides MC. Comparison of Acute Stroke Preparedness Strategies to Decrease Emergency Department Arrival Time in a Multiethnic Cohort: The Stroke Warning Information and Faster Treatment Study. Stroke. 2015 Jul;46(7):1806-12. doi: 10.1161/STROKEAHA.114.008502. Epub 2015 Jun 11. PMID 26069259
- [Derived] Kerns JM, Heidmann D, Petty M, Prabhakaran S. Optimizing public health strategies for stroke education: need for a controlled trial. Am J Ther. 2011 Jan;18(1):81-90. doi: 10.1097/MJT.0b013e3181e123cd. PMID 20634684